CLINICAL TRIAL: NCT00055809
Title: Phase II Study Of Bevacizumab And PEG Interferon Alpha-2b (PEG Intron) In Patients With Metastatic, Or Unresectable Carcinoid Tumors
Brief Title: Bevacizumab and PEG-Interferon Alfa-2b in Treating Patients With Metastatic or Unresectable Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02519; MDA-ID-02063; N01CM62202 (NIH); CDR0000271225 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Gastrointestinal Carcinoid Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Regional Gastrointestinal Carcinoid Tumor
MeSH Terms: interventions — peginterferon alfa-2b; Bevacizumab

ARMS (2):
- Arm I (bevacizumab) (Experimental): Patients receive bevacizumab IV on day 1.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis
- Arm II (PEG-interferon alfa-2b) (Experimental): Patients receive PEG-interferon alfa-2b SC on days 1, 8, and 15.
  Interventions: Biological: PEG-interferon alfa-2b; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Given SC
  Other Names: PEG-IFN alfa-2b; pegylated interferon alfa-2b; polyethylene glycol IFN-A2b
  Arms: Arm II (PEG-interferon alfa-2b)
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I (bevacizumab)
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This randomized phase II trial is to see if combining bevacizumab with PEG-interferon alfa-2b works in treating patients who have metastatic or unresectable carcinoid tumors. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. PEG-interferon alfa-2b may stop the growth of cancer by stopping blood flow to the tumor. Combining bevacizumab with PEG-interferon alfa-2b may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the progression-free survival rate in patients with metastatic or unresectable carcinoid tumors treated with bevacizumab and PEG-interferon alfa-2b.

II. Determine the tumor response rate (complete and partial) in patients treated with this regimen.

III. Determine the biochemical response rate of patients treated with this regimen.

IV. Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients.

OUTLINE: This is a randomized study. Patients are treated in 2 stages.

Stage I: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive bevacizumab IV on day 1.

Arm II: Patients receive PEG-interferon alfa-2b subcutaneously (SC) on days 1, 8, and 15.

In both arms, courses repeat every 3 weeks. Patients with progressive disease at 9 weeks proceed to stage II. All other patients proceed to stage II after 18 weeks on stage I.

Stage II: Patients receive bevacizumab IV on day 1 and PEG-interferon alfa-2b SC once weekly. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) and remain in CR for 2 additional courses come off study. Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoid tumor

  * Metastatic or unresectable local-regional disease
* Measurable disease
* No osseous metastasis as the only site of disease
* No history or clinical evidence of CNS disease (e.g., primary brain tumor or any brain metastasis)
* Performance status - Zubrod 0-2
* Performance status - Karnofsky 70-100%
* At least 12 weeks
* See Immunologic
* Absolute granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8 g/dL
* No bleeding diathesis or coagulopathy
* No hemoglobinopathies (e.g., thalassemia) or any other cause of hemolytic anemia
* Bilirubin < 1.5 mg/dL
* INR < 1.5 (if receiving warfarin)
* No evidence of decompensated liver disease (e.g., ascites, bleeding varices, or spontaneous encephalopathy)
* Creatinine < 1.5 mg/dL
* No baseline proteinuria

  * Patients with proteinuria (≥ 2+ or ≥ 100 mg/dL on urinalysis) are allowed provided 24-hour urinary protein is < 500 mg
* No New York Heart Association grade II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No clinically significant peripheral vascular disease
* No history of stroke
* None of the following within the past 6 months:

  * Uncontrolled hypertension
  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* No chronic pulmonary disease (e.g., chronic obstructive pulmonary disease)
* No documented pulmonary hypertension
* None of the following immunologically mediated diseases:

  * Inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
  * Rheumatoid arthritis
  * Idiopathic thrombocytopenia purpura
  * Systemic lupus erythematosus
  * Autoimmune hemolytic anemia
  * Scleroderma
  * Severe psoriasis
* No serious concurrent infections
* No active infection requiring parental antibiotics on day 0
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No known hypersensitivity to interferon alfa or to any excipient or vehicle included in its formulation or delivery system
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant traumatic injury within the past 4 weeks
* No preexisting thyroid abnormality for which thyroid function can not be normalized by medication
* No concurrent nonmalignant uncontrolled medical illness or one whose control may be jeopardized by the complications of this study therapy
* No uncontrolled psychiatric disorder
* No psychiatric disorders that would preclude study compliance
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No serious nonhealing wound ulcer or bone fracture
* No seizures not controlled with standard medical therapy
* Prior immunotherapy allowed

  * No prior interferon
* No concurrent immunotherapy
* At least 4 weeks since prior chemotherapy, including radiosensitizers
* No more than 1 prior chemotherapy regimen, including radiosensitizers
* No concurrent chemotherapy
* At least 4 weeks since prior radiotherapy

  * Prior radiotherapy must not have contained the single evaluable lesion of this study in a radiation field
* No concurrent radiotherapy
* At least 4 weeks since prior major surgery or open biopsy (1 week for minor surgery) and recovered
* No concurrent or recent full-dose anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting, permanent indwelling IV catheters)
* No concurrent chronic daily aspirin (more than 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-01; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Tumor response rate (CR + PR) as measured by RECIST criteria | Up to 4 years

SECONDARY OUTCOMES:
Progression free survival | From the time of initial treatment to the time of PD or death, assessed up to 4 years
Biochemical response rate measured after treatment | Up to 4 years
Toxicity graded according to CTC v3.0 criteria for adverse outcomes | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States